CLINICAL TRIAL: NCT03455296
Title: Fluid Management Guided With Lactate Clearance Versus Central Venous Oxygen Saturation Monitoring in Surgical Patients in Intensive Care Unit.
Brief Title: Fluid Management Surgical Patients in Intensive Care Unit.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Hepatology & Tropical Medicine Research Institute (Other Government)
Responsible Party: Principal Investigator, ICU, Consultant of Intensive care medicine, Ph D, National Hepatology & Tropical Medicine Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Lactate
Record Dates: First submitted 2018-01-03; First posted 2018-03-06 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Post Operative Fluid Management
MeSH Terms: interventions — Fluid Therapy; Crystalloid Solutions; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- central venous oxygen saturation ScVO2 normalization (Active Comparator): Fluid therapy is initiated with maintenance fluid (Ringer or Ringer acetate) plus replacement with crystalloids (Ringer, Ringer acetate or saline 0.9%) 500ml / 30 min. guided by ScVO2with target value ≥ 70%
  Interventions: Other: fluid therapy; crystalloid
- Lactate clearance (Active Comparator): Fluid therapy is initiated with maintenance fluid (Ringer or Ringer acetate) plus replacement with crystalloids 500ml / 30 min. guided by lactate clearance (LCR) with target value ≤ 2mmol/L (or decline ≥ 10%) by the end of the study
  Interventions: Other: fluid therapy; crystalloid

INTERVENTIONS:
Other: fluid therapy; crystalloid — maintenance fluid e.g. Ringer or Ringer acetate plus replacement fluid with crystalloids e.g. Ringer,or Ringer acetate or saline 0.9%, 500ml / 30 min. guided by ScVO2 with target value ≥ 70% versus lactate clearance (LCR) with target value ≤ 2mmol/L (or decline ≥ 10%) by the end of the study in group A & group B respectively. Maintenance fluid without replacement will be initiated if ScVO2 or lactate value normalized.
  Other Names: Ringeror Ringer acetate or saline 0.9%

SUMMARY:
The aim of this study is to evaluate the efficacy of lactate clearance (LCR) versus central venous oxygen saturation (ScVO2) to guide fluid management for post-operative patients in the intensive care unit (ICU).

DETAILED DESCRIPTION:
Sixty patients will be randomly assigned in a 1:1 manner into two groups; (group A= thirty patients = ScVO2) & (group B = thirty patients =lactate clearance). Fluid therapy will be initiated in each group with maintenance in the form of crystalloid e.g. Ringer or Ringer acetate (in a dose of 30-35 ml/Kg/day) plus replacement with crystalloid e.g. Ringer, Ringer acetate or saline 0.9%, 500 ml over 10-30 min. that will be administered in boluses [7] guided by ScVO2with target value ≥ 70% versus lactate clearance (LCR) with target value ≤ 2mmol/L (or decline ≥ 10%) by the end of the study in group A & group B respectively with close regular clinical monitoring/30min., CVP limits 12-16 cmH2O & mean arterial pressure (MAP) 65-90mmHg. Maintenance fluid without replacement will be initiated alone if ScVO2 or lactate value normalized or are normal from the start.

All demographic data will be obtained including the patients' age, sex, body mass index (BMI), associated co-morbidities (diabetes mellitus &hypertension), Sequential Organ Failure Assessment (SOFA) on admission & discharge from ICU, duration of surgery, the type of surgery, the amount of blood loss intraoperative, the amount of blood transfused intraoperative, the need&the amount of blood transfusion postoperative & will be recorded.

Follow-up hemodynamics including the heart rate, mean arterial pressure (MAP), CVP, arterial oxygen saturation (SaO2), urine volume, fluid balance, blood gases (base excess, PH), hypoxic index (PaO2/FIO2 ratio) & total fluid infused as a baseline then followed as required. Monitoring of either lactate level or ScVO2 on admission followed and recorded at regular intervals during treatment on 0, 2, 6, 12, 24 & 48hours.

Laboratory investigations including the complete blood profile, prothrombin time, liver functions, serum creatinine & serum electrolytes will be assessed at randomization as a baseline & then will be recorded as required. Postoperative medical or surgical morbidities will be followed during ICU & hospital stay e.g. weight gain, impairment of hypoxic index (P/F ratio), pulmonary edema, pleural effusion, need for mechanical ventilation, paralytic ileus, renal impairment& intra-abdominal bleeding.28-day mortality will be asked for & followed by calling the telephone number of the patient or one of his/her first-degree relatives.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are admitted to the intensive care unit of National Hepatology & Tropical Medicine Research Institute (NHTMRI) post intra-abdominal surgical intervention.

Exclusion Criteria:

* Patients will be excluded from the study if they have severe liver impairment (child-Pugh C15), septic shock or hemodynamic instability requiring high dose circulatory support e.g. > 2ug/min noradrenaline as it will impair lactate clearance &/or central venous oxygen saturation normalization, advanced heart failure, central venous pressure (CVP) ≥ 18cmH2O as it will limit fluid therapy, severe hypothermia (< 28◦ C) as it will induce lactate production.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
ICU stay | 2-5 days
  Length of stay in days
medical complications | 2-5 days
  notice any medical complications e.g.infections, pulmonary edema, pleural effusion, need mechanical ventilation, renal impairment
surgical complications | 2-5 days
  notice any surgical complications e.g. wound dehisence, intrabdominal bleeding, ileus

SECONDARY OUTCOMES:
cost of each method | within 48 hours
  cost for fluids given & the method used ScVO2 or Lactate measurements
hospital stay | 2-5 days
  length of stay
mortality | 28 day
  28 day mortality

CONTACTS AND LOCATIONS:
Locations (1):
- NHTMRI, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR, Analytic Code